CLINICAL TRIAL: NCT06858150
Title: Survey on Needle Depth and Angle at Jianzhongshu Acupoint With Ultrasound Guidance Targeting the Levator Scapulae Attachment
Brief Title: Survey on Needle Depth and Angle at Jianzhongshu Acupoint Under Ultrasound Guidance
Status: Completed | Type: Observational
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Doctor of Philosophy, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: 3336/DHYD-HDDD
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Anatomy of Jianzhongshu Acupoint and Levator Scapulae Attachment
Keywords: Ultrasound Guidance; Needle Depth; Needle Angle; Levator Scapulae; Jianzhongshu acupoint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound-Guided Needle Depth and Angle Measurement — This study utilizes ultrasound imaging to measure the needle insertion depth at Jianzhongshu (SI15) and an electronic goniometer to assess insertion angles. The aim is to collect anatomical reference data for acupuncture needling precision, focusing on the relationship between SI15 and the insertion point of the levator scapulae muscle. This is an observational study designed to collect anatomical reference data for acupuncture needling, without evaluating therapeutic effects.

SUMMARY:
The levator scapulae muscle is commonly involved in chronic neck and shoulder pain, with trigger points often located at its insertion on the superior angle of the scapula. Jianzhongshu (SI15) has been identified as a corresponding acupuncture point.

Ultrasound imaging enhances the accuracy and safety of acupuncture by providing real-time visualization of anatomical structures, while electronic goniometry allows precise measurement of needle insertion angles.

This study aims to investigate the depth and angles of needle insertion at SI15 using ultrasound and electronic goniometry. The findings will provide essential anatomical reference data for clinical applications, particularly in acupuncture treatment for neck and shoulder pain.

DETAILED DESCRIPTION:
The levator scapulae muscle is one of the most common muscles involved in chronic neck and shoulder pain. Acupuncture has been widely recognized as an effective and safe treatment for neck pain, with trigger point acupuncture showing significant potential in pain management. In clinical practice, trigger points are often identified at the origin or insertion of the affected muscle. For the levator scapulae, one notable trigger point is located at its insertion point on the superior angle of the scapula. Jianzhongshu (SI15) has been identified as a potential acupuncture point corresponding to this trigger point.

This observational study aims to investigate the anatomical relationship between Jianzhongshu (SI15) and the insertion point of the levator scapulae muscle by assessing the depth and angle of needle insertion using ultrasound and electronic goniometry. The study will recruit healthy adult volunteers aged 18 years and older. Ultrasound imaging will be utilized to measure the needle insertion depth from the skin surface to the insertion point of the levator scapulae muscle. Additionally, an electronic goniometer will be used to assess two specific angles of needle insertion: the angle relative to the skin surface and the angle relative to the longitudinal axis of the body.

The primary objective of this study is to provide anatomical data on the needle insertion depth and angles when needling Jianzhongshu (SI15) toward the insertion point of the levator scapulae muscle. This data will serve as an essential reference for clinical applications, particularly in the treatment of neck and shoulder pain associated with the levator scapulae muscle and SI15.

Secondary objectives include assessing individual variations in needle depth and trajectory, as well as analyzing the influence of demographic factors such as age, gender, and BMI on these parameters.

By integrating ultrasound imaging and an electronic goniometer, this study aims to improve the accuracy and safety of acupuncture needling at SI15. The findings will contribute to a deeper understanding of acupuncture techniques and provide essential reference data for clinical practice, particularly in the management of neck and shoulder pain related to the levator scapulae muscle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 and older
* Ability to understand and consent to participation

Exclusion Criteria:

* Severe chronic diseases or immunocompromised conditions
* Severe exhaustion or widespread infection
* Local infections or wounds at needling sites
* History of surgery or trauma in the target area
* Pregnant or breastfeeding individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers without known musculoskeletal disorders, aged 18 and older, who are eligible for ultrasound-guided acupuncture. Participants are recruited from the community and screened for inclusion and exclusion criteria before enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Needle Depth at Jianzhongshu | During the procedure
  Measurement of needle depth from skin surface to the midpoint of the levator scapulae's distal attachment using ultrasound.
Needle Angle at Jianzhongshu | During the procedure
  Measurement of needle angle relative to the skin surface and spine using an electronic goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Center HCMC - Branch no.3, Ho Chi Minh, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Park JJ, Akazawa M, Ahn J, Beckman-Harned S, Lin FC, Lee K, Fine J, Davis RT, Langevin H. Acupuncture sensation during ultrasound guided acupuncture needling. Acupunct Med. 2011 Dec;29(4):257-65. doi: 10.1136/aim.2010.003616. Epub 2011 Jun 4. PMID 21642648
- [Background] Liang YS, Chen LY, Cui YY, Du CX, Xu YX, Yin LH. Ultrasound-guided acupotomy for trigger finger: a systematic review and meta-analysis. J Orthop Surg Res. 2023 Sep 13;18(1):678. doi: 10.1186/s13018-023-04127-3. PMID 37705066
- [Background] Kwok G, Cohen M, Cosic I. Mapping acupuncture points using multi channel device. Australas Phys Eng Sci Med. 1998 Jun;21(2):68-72. PMID 9745792
- [Background] Mense S. Muscle pain: mechanisms and clinical significance. Dtsch Arztebl Int. 2008 Mar;105(12):214-9. doi: 10.3238/artzebl.2008.0214. Epub 2008 Mar 21. PMID 19629211
- [Background] Itoh K, Katsumi Y, Hirota S, Kitakoji H. Randomised trial of trigger point acupuncture compared with other acupuncture for treatment of chronic neck pain. Complement Ther Med. 2007 Sep;15(3):172-9. doi: 10.1016/j.ctim.2006.05.003. Epub 2006 Jul 10. PMID 17709062
- [Background] Liu L, Skinner MA, McDonough SM, Baxter GD. Traditional Chinese Medicine acupuncture and myofascial trigger needling: The same stimulation points? Complement Ther Med. 2016 Jun;26:28-32. doi: 10.1016/j.ctim.2016.02.013. Epub 2016 Feb 22. PMID 27261978
- [Background] Witt CM, Jena S, Brinkhaus B, Liecker B, Wegscheider K, Willich SN. Acupuncture for patients with chronic neck pain. Pain. 2006 Nov;125(1-2):98-106. doi: 10.1016/j.pain.2006.05.013. Epub 2006 Jun 14. PMID 16781068
- [Background] Vas J, Perea-Milla E, Mendez C, Sanchez Navarro C, Leon Rubio JM, Brioso M, Garcia Obrero I. Efficacy and safety of acupuncture for chronic uncomplicated neck pain: a randomised controlled study. Pain. 2006 Dec 15;126(1-3):245-55. doi: 10.1016/j.pain.2006.07.002. Epub 2006 Aug 23. PMID 16934402
- [Background] Andersen LL, Hansen K, Mortensen OS, Zebis MK. Prevalence and anatomical location of muscle tenderness in adults with nonspecific neck/shoulder pain. BMC Musculoskelet Disord. 2011 Jul 22;12:169. doi: 10.1186/1471-2474-12-169. PMID 21777478